CLINICAL TRIAL: NCT07145996
Title: AI-Enhanced Telerehabilitation Program Using Automated Video Analysis and Personalized Feedback on Pain, Disability, Mobility, Endurance, for Chronic Non-Specific Low Back Pain in College Students: A Randomized Controlled Trial
Brief Title: AI-Enhanced Telerehabilitation Program Using Automated Video Analysis and Personalized Feedback on Pain, Disability, Mobility, Endurance, for Chronic Non-Specific Low Back Pain in College Students.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Collaborators: Galgotias University (Unknown)
Responsible Party: Principal Investigator, faizan kashoo, PT, PhD Scholar, Majmaah University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GALGOTIASUNIVERSITY
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Non Specific Low Back Pain
Keywords: back pain; exercise; young adults; artificial intelligence
MeSH Terms: conditions — Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: This three-arm parallel RCT uses single-blind design to evaluate AI-enhanced telerehabilitation for chronic low back pain in college students. Participants are randomized to: (1) AI-Enhanced Telerehabilitation with computer vision technology (MediaPipe Pose) providing real-time movement analysis and automated feedback via webcam, plus physiotherapist teleconsultations; (2) Standard Telerehabilitation with pre-recorded videos and periodic therapist sessions; or (3) Usual Care control. The AI system tracks exercise performance, counts repetitions, corrects posture, and enables personalized guidance. Primary outcomes include pain, disability, mobility, and trunk endurance over 6 weeks with 3-month follow-up. This addresses the research gap in AI-enhanced remote rehabilitation for young adults.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors evaluating primary endpoints (pain, disability, mobility, trunk endurance) are blinded to group allocation to prevent measurement bias. Independent research assistants conducting assessments remain unaware of participants' intervention assignments.
  Participants cannot be blinded due to intervention nature - they know whether receiving AI-enhanced telerehabilitation, standard telerehabilitation, or usual care. Physiotherapists delivering interventions cannot be blinded as they provide group-specific treatments.
  Data analysts remain blinded to group codes during statistical analysis until primary analyses complete. Principal investigator maintains randomization knowledge for safety monitoring but doesn't participate in outcome measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AI-Enhanced Telerehabilitation (Experimental): Participants receive personalized exercise programs delivered through a custom telerehabilitation platform incorporating AI-based movement analysis using Google MediaPipe Pose computer vision technology. The system monitors exercise performance through participants' webcams or smartphones, providing real-time feedback on form, automatically counting repetitions, measuring hold times, and flagging technique errors. AI-generated performance data is reviewed by physiotherapists who provide personalized corrective guidance through scheduled video consultations. Exercises focus on flexibility, core stability, and functional strength targeting chronic non-specific low back pain. The intervention combines objective AI monitoring with human therapeutic guidance to optimize exercise adherence and technique.
  Interventions: Other: AI Based Exercises
- Exercise-Only Telerehabilitation (Active Comparator): Participants receive structured exercise programs delivered via pre-recorded video instructions without AI monitoring or automated feedback. This represents current standard telerehabilitation practice, with periodic physiotherapist consultations conducted through video conferencing sessions. Exercise programs include the same flexibility, core stability, and functional strength components as the AI-enhanced group, but without objective movement analysis or real-time form correction. Therapists rely on visual observation during video sessions and participant self-reports to monitor progress and provide guidance. This arm serves as an active control to isolate the specific effects of AI-enhanced monitoring and feedback.
  Interventions: Other: Standard Telerehabilitation
- Usual Care (No Intervention): This control intervention represents standard medical care typically provided to college students with chronic non-specific low back pain. Participants receive general advice on activity modification, recommendations for over-the-counter pain medications (NSAIDs, acetaminophen), basic exercise suggestions, and routine follow-up appointments as clinically indicated. No structured exercise program, telerehabilitation platform, or specialized physiotherapy intervention is provided. Participants may seek additional healthcare services as they normally would, including visits to primary care physicians, specialists, or other healthcare providers. This arm serves as a control group to evaluate the effectiveness of both telerehabilitation interventions against current standard medical management practices.

INTERVENTIONS:
Other: AI Based Exercises — This intervention combines structured exercise therapy with artificial intelligence-powered movement analysis using Google MediaPipe Pose technology. Participants perform prescribed exercises (flexibility, core stability, functional strength) while a computer vision system analyzes their movements through standard webcam or smartphone cameras. The AI provides real-time feedback on exercise form, automatically counts repetitions, measures hold times, and flags technique errors. Physiotherapists review AI-generated performance data and provide personalized corrective guidance through scheduled video consultations. The platform delivers 8-week progressive exercise programs specifically designed for chronic non-specific low back pain, integrating objective movement monitoring with human therapeutic oversight to optimize adherence and clinical outcomes.
  Arms: AI-Enhanced Telerehabilitation
Other: Standard Telerehabilitation — This intervention delivers structured exercise therapy through pre-recorded video instructions without AI monitoring or automated feedback. Participants receive the same exercise components as the AI-enhanced group (flexibility, core stability, functional strength) but rely on video demonstrations and written instructions for proper technique. Physiotherapists conduct periodic consultations via video conferencing to monitor progress, provide guidance, and adjust exercise programs based on visual observation and participant self-reports. The 8-week progressive program represents current standard telerehabilitation practice for chronic non-specific low back pain, serving as an active comparator to isolate the specific effects of AI-enhanced movement analysis and real-time feedback systems.
  Arms: Exercise-Only Telerehabilitation

SUMMARY:
This study tests whether an artificial intelligence (AI)-enhanced telerehabilitation program can effectively treat chronic non-specific low back pain in college students.

Low back pain affects 40-52% of university students due to prolonged sitting during lectures and study sessions, poor posture from laptop use, and lack of physical activity. While exercise therapy is the recommended treatment, many students cannot access traditional physiotherapy due to cost, scheduling conflicts, and location barriers.

This randomized controlled trial compares three treatment approaches: (1) AI-enhanced telerehabilitation with automated video analysis and personalized feedback, (2) standard telerehabilitation with video instructions only, and (3) usual care. The AI system uses computer vision technology (Google MediaPipe Pose) to analyze exercise videos through a standard webcam or smartphone, automatically tracking joint movements, counting repetitions, and providing real-time feedback on exercise form.

College students with chronic low back pain (lasting more than 3 months) will be randomly assigned to one of the three groups. The AI-enhanced group will receive personalized exercise programs delivered remotely, with the AI system monitoring their performance and physiotherapists providing guidance through video consultations.

The study will measure changes in pain levels, disability, physical function, trunk muscle endurance, and quality of life over 8 weeks of treatment and 3 months of follow-up. Researchers will also evaluate how well participants stick to their exercise programs and how easy the technology is to use.

This research aims to determine if AI technology can make remote physiotherapy more effective and accessible for college students, potentially transforming how young adults receive treatment for back pain and improving their long-term health outcomes.

DETAILED DESCRIPTION:
Chronic non-specific low back pain (CNSLBP) has emerged as a significant health concern among college students, with international studies reporting prevalence rates between 40-52%. This high incidence is attributed to the modern academic environment, characterized by prolonged static postures during lectures and study sessions, extensive use of laptops and handheld devices leading to poor trunk alignment, and generally low levels of structured physical activity resulting in deconditioning of core and postural muscles.

The impact of CNSLBP in college students extends beyond physical discomfort, affecting academic performance, causing absenteeism, limiting recreational participation, and potentially leading to persistent pain patterns in adulthood. Current evidence-based management guidelines recommend multidisciplinary approaches emphasizing structured exercise therapy, self-management education, and postural retraining, with particular focus on flexibility, core stability, and functional strength exercises.

However, significant barriers prevent college students from accessing optimal care. These include logistical challenges such as academic scheduling conflicts, economic constraints related to repeated physiotherapy visits, and geographical accessibility issues. Consequently, many students resort to unsupervised home exercise programs that, while cost-effective and flexible, lack real-time monitoring and professional guidance, often resulting in incorrect technique, poor adherence, and suboptimal outcomes.

TECHNOLOGICAL INNOVATION

Recent advances in artificial intelligence (AI) and computer vision technology offer promising solutions to bridge this care gap. Markerless motion capture systems, particularly Google's MediaPipe Pose and OpenPose, can analyze human movement using standard cameras to identify skeletal landmarks, track joint angles, assess posture, and detect movement deviations in real-time. These systems demonstrate approximately 85% accuracy for gross movement tracking and exercise repetition counting, making them suitable for clinical rehabilitation applications.

When integrated into telerehabilitation platforms, AI-driven video analysis provides dual benefits: enhancing remote care quality by supplying therapists with quantitative performance feedback, and enabling patients to receive immediate automated correction cues, thereby improving engagement and self-efficacy.

STUDY DESIGN AND METHODOLOGY

This single-blind, three-arm parallel-group randomized controlled trial will compare the effectiveness of AI-enhanced telerehabilitation versus standard telerehabilitation and usual care in college students with CNSLBP. The study design addresses a critical research gap, as no published randomized controlled trials have specifically examined AI-enhanced telerehabilitation in this population.

INTERVENTION GROUPS

Group 1: AI-Enhanced Telerehabilitation Participants will receive personalized exercise programs delivered through a custom platform incorporating AI-based movement analysis. The system uses computer vision algorithms to monitor exercise performance through participants' webcams or smartphones, providing real-time feedback on form, automatically counting repetitions, measuring hold times, and flagging technique errors. Physiotherapists will review AI-generated performance data and provide personalized guidance through scheduled video consultations.

Group 2: Standard Telerehabilitation Participants will receive exercise programs via video instructions without AI monitoring or personalized feedback. This group represents current telerehabilitation practice, relying on pre-recorded exercise videos and periodic therapist consultations without objective movement analysis.

Group 3: Usual Care Control Participants will receive standard medical care as typically provided for CNSLBP, which may include general advice on activity modification, over-the-counter pain medications, and basic exercise recommendations without structured supervision.

PARTICIPANT SELECTION

The study will recruit college students aged 18-25 years with chronic non-specific low back pain (duration >3 months) from university health services and campus recruitment. Inclusion criteria ensure participants have clinically significant symptoms warranting intervention, while exclusion criteria eliminate cases with specific pathologies requiring specialized medical management.

OUTCOME MEASURES

Primary outcomes include pain intensity measured using the Numerical Rating Scale (NRS), functional disability assessed with the Roland-Morris Disability Questionnaire (RMDQ), functional mobility evaluated through the Timed Up and Go (TUG) test, and trunk muscular endurance measured via the prone plank test. These validated instruments are sensitive to clinical changes in low back pain populations.

Secondary outcomes encompass adherence rates to prescribed exercises, platform usability assessed through standardized questionnaires, quality of life measures, healthcare utilization patterns, and long-term follow-up assessments at 3 months post-intervention.

STATISTICAL ANALYSIS

The study will employ intention-to-treat analysis as the primary approach, with per-protocol analysis as secondary. Power calculations indicate adequate sample size to detect clinically meaningful differences between groups. Mixed-effects models will account for repeated measurements and potential confounding variables.

EXPECTED OUTCOMES AND SIGNIFICANCE

This research aims to establish whether AI-enhanced telerehabilitation can provide superior clinical outcomes compared to standard approaches while maintaining high usability and adherence rates. The findings have potential to inform university health services, influence physiotherapy practice guidelines, and support broader integration of AI technology into telehealth delivery.

The study aligns with the World Health Organization's Global Strategy on Digital Health 2020-2025, which encourages leveraging digital innovation to improve healthcare accessibility and equity. By focusing on a tech-savvy demographic experiencing significant barriers to traditional care, this research addresses both immediate clinical needs and broader healthcare delivery challenges.

INNOVATION AND FUTURE IMPLICATIONS

This study represents a pioneering application of AI technology in rehabilitation for young adults, potentially establishing a scalable model for remote physiotherapy delivery. The integration of objective movement analysis with personalized professional guidance offers a novel approach that maintains therapeutic relationships while leveraging technological capabilities for enhanced monitoring and feedback.

The research contributes to the growing body of evidence supporting digital health interventions while specifically addressing the unique needs and circumstances of college students with chronic low back pain. Success could lead to broader implementation across university health systems and expansion to other musculoskeletal conditions and age groups.

QUALITY ASSURANCE

The study incorporates rigorous methodological standards including randomization procedures, blinding where possible, validated outcome measures, standardized intervention protocols, and comprehensive statistical analysis plans. Regular monitoring ensures protocol adherence and participant safety throughout the study period.

ELIGIBILITY:
Inclusion Criteria

* Age 18-30 years, currently enrolled in undergraduate or postgraduate study.
* Diagnosis of non-specific LBP for at least 3 months.
* Baseline pain intensity between 3 and 7 (NRS).
* Ability and willingness to perform prescribed exercises and participate in video conferencing.
* Access to suitable device and reliable internet.
* Informed consent obtained. Exclusion Criteria
* Specific causes of LBP (e.g., fracture, tumor, infection, inflammatory disease).
* Recent spinal surgery or confirmed disc herniation (within past year).
* Neurological deficits or severe comorbid conditions contraindicating exercise.
* Pregnancy or current participation in another structured LBP program.
* BMI ≥ 35 kg/m² (could impair AI pose detection).
* Inability to understand English instructions or complete measures.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | From enrollment to the end of treatment at 6 week and 3 months
  A unidimensional measure of pain intensity in which participants rate their average low back pain over the past week on an 11-point scale from 0 ("no pain") to 10 ("worst imaginable pain"). The NRS is valid, reliable, and sensitive to clinical change in chronic low back pain populations.

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire (RMDQ) | From enrollment to the end of treatment at 6 weeks and 3 months
  A 24-item self-report inventory assessing functional disability due to low back pain. Each affirmative response (e.g., "I stay at home most of the time because of my back") scores one point; total scores range from 0 (no disability) to 24 (maximum disability). The RMDQ demonstrates excellent test-retest reliability and responsiveness in non-specific low back pain.
Timed Up and Go (TUG) Test | From enrollment to the end of treatment at 6 weeks and 3 months
  An objective measure of basic functional mobility and fall risk. Participants rise from a seated position, walk 3 meters at a comfortable pace, turn, return, and sit down; time to completion is recorded in seconds. The TUG test is reliable, valid, and sensitive to changes in dynamic balance and gait speed in musculoskeletal populations.
Prone Plank Test | From enrollment to the end of treatment at 6 weeks and 3 months
  An assessment of trunk muscular endurance. Participants assume a prone forearm plank position with elbows under shoulders and body in a straight line from head to heels and hold as long as possible; duration is recorded in seconds. The prone plank test correlates with core stability and functional performance in chronic low back pain.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code